CLINICAL TRIAL: NCT04257214
Title: Identifying Optimal Psychosocial Interventions for Patients Receiving Office-Based Buprenorphine
Brief Title: Therapy and Peer Support for Patients Taking Medication for Opioid Use Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philadelphia College of Osteopathic Medicine (Other)
Collaborators: Boston University (Other); Patient-Centered Outcomes Research Institute (Other); Public Health Management Corporation (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: OBOT-2018C2-13158
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Opioid Use Disorder
Keywords: Opioid Use; Buprenorphine; Psychosocial Treatment; Medication Assisted Treatment; Cognitive Behavioral Therapy; Peer Support; Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Treatment as usual (No Intervention): Those randomized to treatment as usual will receive standard treatment from one of four FQHC sites.
- Office based CBT (Active Comparator): Those randomized to Cognitive Behavioral Treatment will receive cognitive behavioral treatment (CBT) along with standard treatment from the FQHC.
  Interventions: Behavioral: Psychosocial treatment
- CRS/CPS (Active Comparator): Those randomized to certified recovery specialist(CRS)/peer support specialist(CPS) will receive a CRS/CPS along with standard treatment from the FQHC.
  Interventions: Behavioral: Psychosocial treatment
- CBT+CRS/CPS (Active Comparator): Those randomized to MAT+ office-based CBT will receive office-based buprenorphine treatment along with office-based CBT and a CRS.
  Interventions: Behavioral: Psychosocial treatment

INTERVENTIONS:
Behavioral: Psychosocial treatment — Participants randomly assigned to one of four psychosocial treatment conditions including cognitive behavioral therapy and a certified recovery specialist.
  Arms: CBT+CRS/CPS; CRS/CPS; Office based CBT

SUMMARY:
Current clinical guidelines for medication assisted treatment (MAT) of opioid use disorder (OUD) recommend that treatment include a psychosocial component to help address psychological factors related to addiction. However, a knowledge gap exists regarding the most effective forms of psychosocial intervention and what interventions are most effective for different types of patients. This gap represents a significant barrier to the widespread implementation of effective office-based opioid treatment (OBOT) with buprenorphine, which is important to improving opioid treatment and responding to the critical needs of individuals living with OUD. The overarching goal of this patient-centered research is to address the diverse needs and preferences of OUD patients in regards to psychosocial approaches and to overcome the "one-size-fits-all" strategies that are typically used to treat OUD. Importantly, investigators arrived at this goal, in part, through collaboration and consultation with former patients who have received different types of treatments for OUD. In this manner, patients provided important insight to inform the selection of interventions to be evaluated, patient characteristics that may differentially impact the effects of the interventions, and the patient outcomes to be examined.

DETAILED DESCRIPTION:
The study will evaluate the comparative effectiveness of two psychosocial approaches, Cognitive Behavioral Therapy and peer support through the use of Certified Recovery Specialists (CRS's)/ Certified Peer Specialists (CPS's) provided within the context of office-based buprenorphine treatment. Patients will be randomly assigned to receive either (1) standard Medication Management (MM) as typically provided at the site, (2) MM with office-based CBT, (3) MM with CRS/CPS, and (4) MM with both CBT and CRS/CPS. In MM, patients will be seen by providers at least weekly until stable, and stabilized patients will then be seen by the provider on a monthly basis. If a patient needs a higher level of care, they will be referred to appropriate specialty treatment to ensure their safety. In the CBT study arms, CBT will be provided through 12 individual manualized sessions scheduled to coincide with patients' MM appointments when possible. As outlined by the National Institute on Drug Abuse (NIDA), sessions will cover standard CBT topics and include exercises and homework. Meta-analyses and reviews have concluded that CBT is an effective treatment across a range of SUDs and has helped to enhance treatment retention, improve medication adherence, and address ancillary problems. In the CRS/CPS study arms, CRS's/CPS's will meet with clients following their first OBOT session to assist them in accessing community resources and overcoming treatment barriers, and provide ongoing patient navigation services to promote attendance at OBOT appointments. These appointments will occur either in-person or over the phone and all meetings will be tracked by the CRS/CPS. Studies indicate that peer-delivered services for individuals with mental health disorders are effective in engaging "difficult-to-reach" individuals and improving multidimensional outcomes. In the combined CBT/CRS study arm, clients will receive the individual CBT sessions and be assigned to a CRS/CPS.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Be deemed eligible for buprenorphine treatment for OUD by the FQHC treatment provider and agree to engage in this treatment;
* Not require an inpatient level of care as determined by the healthcare provider;
* Be capable of providing valid contact information and informed consent; and
* Permit the research team to use and disclose their protected health information (PHI).

Exclusion Criteria:

Individuals who are intoxicated, cognitively impaired, or psychiatrically unstable at baseline will not be included; however, they may subsequently be included if the disqualifying condition subsides.

DSM 5 criteria for OUD include:

* Taking opioids in larger amounts or longer than intended;
* Failed efforts to quit or cut back;
* Spending a lot of time obtaining the opioid;
* Craving or urges to use;
* Repeated inability to carry out major work, school, or home obligations;
* Continued use despite persistent or recurring interpersonal problems worsened by opioid use;
* Stopping or reducing important social, recreational activities due to opioid use;
* Recurrent use of opioids in physically hazardous situations;
* Continued opioid use despite knowledge of having a persistent or recurrent physical or psychological problem that is likely to have been caused or exacerbated by the substance;
* Tolerance; and
* Withdrawal. Moderate OUD severity is denoted by the presence of 4 or 5 of these symptoms and severe OUD is denoted by 6 or more symptoms. Patients will be excluded from the study if their SUD is primarily for a different substance, or their co-morbid psychiatric needs indicate enhanced needs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Urinalysis-confirmed opioid use | Through 12 months post-study entry
  Participants will provide a urine specimen at baseline and 3, 6, 9, and 12-month assessments. We will use the CLIA Waived® 14-Panel Drug Test Cup and fentanyl test strip for opioids, buprenorphine, methadone, oxycodone, THC, cocaine, amphetamines, PCP, methamphetamine, benzodiazepines, and barbiturates, and MDMA. The urine sample will be delivered under the supervision of the RA who will use standard procedures to detect tampering and dilution.

SECONDARY OUTCOMES:
Retention in Office-Based Buprenorphine Treatment | Through 12 months post-study entry
  Information from the electronic health record (EHR) will be used to determine engagement in OBOT. We will obtain data from the EHR reflecting OBOT-related data including appointments attended, prescription refill information, and service dates. A patient will be identified as having dropped out of OBOT when 30 days without current buprenorphine prescription or 30 days without meeting with provider have passed.
Quality of life assessment | Through 12 months post-study entry
  Quality of life will be measured using the Short Form-36 (SF-36). The SF-36 is a self-report inventory that assesses eight dimensions of physical and mental health-related quality of life. The SF-36 has been shown to have high reliability and validity. The SF-36 individual item scores are recoded to values from 0-100. Items in the same scale are then averaged together to create the 8 scale scores. The scales include physical functioning, role limitations die to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health. A higher score indicates a more positive outcome in the scale.
Multidimensional problem severity | Through 12 months post-study entry
  Multidimensional problem severity, a secondary outcome, will be measured using the Addiction Severity Index-Lite (ASI-Lite). The ASI-Lite is a reliable and valid multidimensional assessment that provides composite scores reflecting current problem severity in the medical, employment, alcohol, drug, legal, family/social, and psychiatric areas. The Addiction Severity Index-Lite yields problem severity scores for the following psychosocial dimensions: drug, alcohol, employment, medical, legal, psychiatric, and family/social. Within each dimension, scores can range from 0 to 1 with higher scores indicating higher problem severity.
Urinalysis-confirmed use from other (non-opioid) drugs | Through 12 months post-study entry
  Results from the CLIAwaived® 14-panel test and fentanyl strip described above for the primary outcome will be used as an indicator of this outcome.
ED utilization | Through 12 months post-study entry
  The Addiction Severity Index-Lite (ASI-Lite) yields problem severity scores for the following psychosocial dimensions: drug, alcohol, employment, medical, legal, psychiatric, and family/social. Within each dimension, scores can range from 0 to 1 with higher scores indicating higher problem severity. The ASI-Lite captures the number of ED visits that the patient experienced during the given timeframe (i.e., past 90 days).
Opioid overdose rates | Through 12 months post-study entry
  The ASI-Lite (see above) captures the number of opioid overdoses that a patient experienced during the given timeframe (i.e., past 90 days). In addition, opioid overdoses will be extracted from the patient's clinical record.
Treatment satisfaction | Through 12 months post-study entry
  Treatment satisfaction will be measured using a subscale from the Client Satisfaction Questionnaire-8. The CSQ-8 measures patient therapeutic engagement in and satisfaction with treatment. Individual scores from the 8 items are added and scores can range from 8-32 with a higher score indicating greater satisfaction.

OTHER OUTCOMES:
Provider outcome: Job satisfaction and stress | Through study completion, an average of 1 year
  We will hold focus groups with all key members of the clinical care team at each Federally Qualified Health Center (FQHC) site following completion of the trial to examine their perceptions about how the study interventions impacted their job-related stress and job satisfaction. The discussion will center on how the different interventions, separately or in combination, influenced the providers.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle R Lent, Ph.D., Principal Investigator — Philadelphia College of Osteopathic Medicine
Locations (5):
- United States (5):
  - AtlantiCare, Atlantic City, New Jersey
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Care Clinic, Philadelphia, Pennsylvania
  - Delaware Valley Community Health, Philadelphia, Pennsylvania
  - Berks Community Health Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kampman K, Jarvis M. American Society of Addiction Medicine (ASAM) National Practice Guideline for the Use of Medications in the Treatment of Addiction Involving Opioid Use. J Addict Med. 2015 Sep-Oct;9(5):358-67. doi: 10.1097/ADM.0000000000000166. PMID 26406300
- [Background] Center for Substance Abuse Treatment. Clinical Guidelines for the Use of Buprenorphine in the Treatment of Opioid Addiction. Rockville (MD): Substance Abuse and Mental Health Services Administration (US); 2004. Report No.: (SMA) 04-3939. Available from http://www.ncbi.nlm.nih.gov/books/NBK64245/ PMID 22514846
- [Background] Davoli M, Amato L, Clark N, Farrell M, Hickman M, Hill S, Magrini N, Poznyak V, Schunemann HJ. The role of Cochrane reviews in informing international guidelines: a case study of using the Grading of Recommendations, Assessment, Development and Evaluation system to develop World Health Organization guidelines for the psychosocially assisted pharmacological treatment of opioid dependence. Addiction. 2015 Jun;110(6):891-8. doi: 10.1111/add.12788. Epub 2014 Dec 10. PMID 25490943
- [Background] Dugosh K, Abraham A, Seymour B, McLoyd K, Chalk M, Festinger D. A Systematic Review on the Use of Psychosocial Interventions in Conjunction With Medications for the Treatment of Opioid Addiction. J Addict Med. 2016 Mar-Apr;10(2):93-103. doi: 10.1097/ADM.0000000000000193. PMID 26808307
- [Background] Schwartz RP. When Added to Opioid Agonist Treatment, Psychosocial Interventions do not Further Reduce the Use of Illicit Opioids: A Comment on Dugosh et al. J Addict Med. 2016 Jul-Aug;10(4):283-5. doi: 10.1097/ADM.0000000000000236. PMID 27471920
- [Background] Department of Health and Human Services. Medication assisted treatment for opioid use disorder (42 CFR Part 8, RIN 0930-AA22). Rockville, MD: Substance Abuse and Mental Health Services Administration.
- [Background] Fiellin DA, Moore BA, Sullivan LE, Becker WC, Pantalon MV, Chawarski MC, Barry DT, O'Connor PG, Schottenfeld RS. Long-term treatment with buprenorphine/naloxone in primary care: results at 2-5 years. Am J Addict. 2008 Mar-Apr;17(2):116-20. doi: 10.1080/10550490701860971. PMID 18393054
- [Background] Alford DP, LaBelle CT, Kretsch N, Bergeron A, Winter M, Botticelli M, Samet JH. Collaborative care of opioid-addicted patients in primary care using buprenorphine: five-year experience. Arch Intern Med. 2011 Mar 14;171(5):425-31. doi: 10.1001/archinternmed.2010.541. PMID 21403039
- [Background] Haddad MS, Zelenev A, Altice FL. Integrating buprenorphine maintenance therapy into federally qualified health centers: real-world substance abuse treatment outcomes. Drug Alcohol Depend. 2013 Jul 1;131(1-2):127-35. doi: 10.1016/j.drugalcdep.2012.12.008. Epub 2013 Jan 17. PMID 23332439
- [Background] Dutra L, Stathopoulou G, Basden SL, Leyro TM, Powers MB, Otto MW. A meta-analytic review of psychosocial interventions for substance use disorders. Am J Psychiatry. 2008 Feb;165(2):179-87. doi: 10.1176/appi.ajp.2007.06111851. Epub 2008 Jan 15. PMID 18198270
- [Background] Amato L, Minozzi S, Davoli M, Vecchi S. Psychosocial and pharmacological treatments versus pharmacological treatments for opioid detoxification. Cochrane Database Syst Rev. 2011 Sep 7;(9):CD005031. doi: 10.1002/14651858.CD005031.pub4. PMID 21901695
- [Background] McHugh RK, Hearon BA, Otto MW. Cognitive behavioral therapy for substance use disorders. Psychiatr Clin North Am. 2010 Sep;33(3):511-25. doi: 10.1016/j.psc.2010.04.012. PMID 20599130
- [Background] Moore BA, Barry DT, Sullivan LE, O'connor PG, Cutter CJ, Schottenfeld RS, Fiellin DA. Counseling and directly observed medication for primary care buprenorphine maintenance: a pilot study. J Addict Med. 2012 Sep;6(3):205-11. doi: 10.1097/ADM.0b013e3182596492. PMID 22614936
- [Background] Fiellin DA, Barry DT, Sullivan LE, Cutter CJ, Moore BA, O'Connor PG, Schottenfeld RS. A randomized trial of cognitive behavioral therapy in primary care-based buprenorphine. Am J Med. 2013 Jan;126(1):74.e11-7. doi: 10.1016/j.amjmed.2012.07.005. PMID 23260506
- [Background] Ling W, Hillhouse M, Ang A, Jenkins J, Fahey J. Comparison of behavioral treatment conditions in buprenorphine maintenance. Addiction. 2013 Oct;108(10):1788-98. doi: 10.1111/add.12266. Epub 2013 Jul 12. PMID 23734858
- [Background] Moore BA, Fiellin DA, Barry DT, Sullivan LE, Chawarski MC, O'Connor PG, Schottenfeld RS. Primary care office-based buprenorphine treatment: comparison of heroin and prescription opioid dependent patients. J Gen Intern Med. 2007 Apr;22(4):527-30. doi: 10.1007/s11606-007-0129-0. PMID 17372805
- [Background] Weiss RD, Potter JS, Fiellin DA, Byrne M, Connery HS, Dickinson W, Gardin J, Griffin ML, Gourevitch MN, Haller DL, Hasson AL, Huang Z, Jacobs P, Kosinski AS, Lindblad R, McCance-Katz EF, Provost SE, Selzer J, Somoza EC, Sonne SC, Ling W. Adjunctive counseling during brief and extended buprenorphine-naloxone treatment for prescription opioid dependence: a 2-phase randomized controlled trial. Arch Gen Psychiatry. 2011 Dec;68(12):1238-46. doi: 10.1001/archgenpsychiatry.2011.121. Epub 2011 Nov 7. PMID 22065255
- [Background] Litz M, Leslie D. The impact of mental health comorbidities on adherence to buprenorphine: A claims based analysis. Am J Addict. 2017 Dec;26(8):859-863. doi: 10.1111/ajad.12644. Epub 2017 Nov 16. PMID 29143483
- [Background] Bassuk EL, Hanson J, Greene RN, Richard M, Laudet A. Peer-Delivered Recovery Support Services for Addictions in the United States: A Systematic Review. J Subst Abuse Treat. 2016 Apr;63:1-9. doi: 10.1016/j.jsat.2016.01.003. Epub 2016 Jan 13. PMID 26882891
- [Background] Reif S, Braude L, Lyman DR, Dougherty RH, Daniels AS, Ghose SS, Salim O, Delphin-Rittmon ME. Peer recovery support for individuals with substance use disorders: assessing the evidence. Psychiatr Serv. 2014 Jul;65(7):853-61. doi: 10.1176/appi.ps.201400047. PMID 24838535
- [Background] Moore BA, Fiellin DA, Cutter CJ, Buono FD, Barry DT, Fiellin LE, O'Connor PG, Schottenfeld RS. Cognitive Behavioral Therapy Improves Treatment Outcomes for Prescription Opioid Users in Primary Care Buprenorphine Treatment. J Subst Abuse Treat. 2016 Dec;71:54-57. doi: 10.1016/j.jsat.2016.08.016. Epub 2016 Sep 2. PMID 27776678
- [Derived] Lent MR, Dugosh KL, Hurstak E, Callahan HR, Mazur K; Greater Philadelphia Opioid Use Disorder Research Group. Prevalence and predictors of suicidality among adults initiating office-based buprenorphine. Addict Sci Clin Pract. 2023 Jun 1;18(1):37. doi: 10.1186/s13722-023-00393-y. PMID 37264472